CLINICAL TRIAL: NCT04240834
Title: Safety and Efficacy of Ticagrelor With Low-dose Aspirin Versus Regular Aspirin in Patients With Acute Coronary Syndrome at High-risk for Ischemia After Percutaneous Coronary Intervention: A Randomized Controlled Study
Brief Title: Ticagrelor With Low-dose Versus Regular Aspirin in Patients With Acute Coronary Syndrome (ACS) at High-Risk for Ischemia After Percutaneous Coronary Intervention
Acronym: LD-ASPIRIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fu Wai Hospital, Beijing, China (Other)
Responsible Party: Principal Investigator, Qian Haiyan, MD, PhD, Fu Wai Hospital, Beijing, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019XK320061
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndrome; Interventional Cardiology
Keywords: ACS; PCI; DAPI; Aspirin; Ticagrelor
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Aspirin; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LD group (Experimental): Low-dose Aspirin(50mg qd) + Ticagrelor( 90mg bid) for 12 months
  Interventions: Drug: Aspirin; Drug: Ticagrelor
- Control group (Active Comparator): Regular Aspirin(75mg qd) + Ticagrelor(90mg bid) for 12 months
  Interventions: Drug: Aspirin; Drug: Ticagrelor

INTERVENTIONS:
Drug: Aspirin — Comparison of 12 months of ticagrelor and low-dose aspirin versus 12 months of standard dual anti-platelet therapy (DAPT)
  Other Names: Acetylsalicylic Acid
Drug: Ticagrelor — Comparison of 12 months of ticagrelor and low-dose aspirin versus 12 months of standard dual anti-platelet therapy (DAPT)
  Other Names: Brilinta/Brilique

SUMMARY:
The present study is aimed to compare the safety and efficacy of Ticagrelor with low-dose Aspirin versus standard dual anti-platelet therapy (DAPT) in patients with acute coronary syndrome (ACS) at high risk for ischemic events after percutaneous coronary intervention (PCI) and stent implantation.

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, blinded-endpoint evaluation, single-center Study. There will be 1220 ACS patients at high risk for ischemic events after successful PCI with implantation of at least one drug eluting stent who will be enrolled in Fuwai Hospital, China. Then those included subjects will be randomized to either Ticagrelor plus low-dose Aspirin (50mg daily, LD group) or Ticagrelor plus regular dose Aspirin (75mg daily, control group) for 12 months. The primary endpoint of the current study is to determine the impact of low-dose Aspirin plus Ticagrelor versus standard DAPT for 12 months on major adverse cardiac and cerebral events (MACCEs), and the secondary endpoint is to determine whether the protocol of low dose Aspirin plus Ticagrelor reduces bleeding events, sufficiently inhibits platelet function, and increases the medication adherence among the included patients. In summary, the present study is to provide new evidence and strategy about the anti-platelet protocol for ACS patients at high risk for ischemia.

ELIGIBILITY:
Inclusion Criteria:

* ACS patients at high risk for ischemic events after successful PCI with implantation of at least one drug eluting stent
* Able and willing to provide informed consent and participate in 12 months follow-up period
* Able to receive DAPT treatment
* Enrollment into the study will require meeting at least one angiographic or clinical inclusion and none of the exclusion criteria.

Clinical inclusion criteria:

1. Family history of premature coronary heart disease (Coronary heart disease in first-degree male relative <55 years old or in first-degree female relative <65 years old)
2. Repeated myocardial infarction
3. Positive serum cardiac troponin I/T
4. Combined with at least one organ/system with atherosclerotic disease (e.g. intracranial or peripheral arteries)
5. Type 2 diabetes mellitus under medication
6. Chronic kidney disease (eGFR<60 mL/min/1.73 m2 or CrCl<60ml/min)

Angiographic Inclusion Criteria:

1. LM lesion requiring stents
2. Proximal LAD lesion(s) requiring stents
3. Bypass grafts lesion(s) requiring stents
4. Overall stent length ≥60 mm
5. History of in-stent thrombosis
6. Bifurcation lesions requiring at least 2 stents
7. Over two vessels lesions requiring stents
8. Calcified target lesion(s) requiring atherectomy
9. The intraoperative occurrence of no-reflow or slow-flow
10. Compressed branch vessels with a diameter of at least 2.0 mm failing to reach flow restoration (at least TIMI 3)

Exclusion Criteria:

* Need for chronic oral anticoagulation
* With cardiomyopathy（HCM/DCM/RCM）
* With severe ventricular arrhythmia requiring ICD implantation
* With chronic respiratory disease (COPD, asthma, chronic bronchitis, pulmonary heart disease)
* With severe infectious disease（active hepatitis B, active hepatitis C, AIDS）
* With hematological disorders（thrombocytopenia, severe anemia, leukaemia）
* With severe liver disease or kidney failure
* With malignant tumor
* With cognitive impairment
* Unable or unwilling to provide informed consent or undergo follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebral events (MACCEs) | 12 months after randomization
  Number of participants with a composite of all-cause mortality, non-fatal myocardial infarction, non-fatal stroke or urgent target vessel revascularization

SECONDARY OUTCOMES:
Bleeding episode (Key secondary endpoint) | 12 months after randomization
  Number of participants with major bleeding(Bleeding Academic Research Consortium (BARC) types ≥3) and/or minor bleeding(Bleeding Academic Research Consortium (BARC) types 0-2)
Platelet function | 12 months after randomization
  Platelet inhibition, blood level and urine level of thromboxaneB2(TXB2)
Medication adherence | 12 months after randomization
Bleeding-related withdrawal | 12 months after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Haiyan Qian, MD, PhD, Principal Investigator — Fuwai Hospital, Beijing, China
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China